CLINICAL TRIAL: NCT02435836
Title: An Open-Label Follow-on Study of the Long-Term Safety of Aripiprazole in Patients With Chronic Schizophrenia
Brief Title: A Follow-on Study of the Long-Term Safety of Aripiprazole in Patients With Chronic Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated when aripiprazole available commercially per protocol
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-97-303
Record Dates: First submitted 2015-04-15; First posted 2015-05-06 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): All subjects began open-label treatment with 30 mg aripiprazole on the first day of participation in the current trial. Once a subject stabilized at the 30 mg per day dose, the investigator could adjust the dose within the range of 10 to 30 mg per day as needed (throughout this long-term trial), to manage AEs.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify

SUMMARY:
The primary objective of the study was to determine the safety of aripiprazole administered long-term in doses ranging from 10 to 30 mg per day as a maintenance therapy in subjects with chronic or first episode of schizophrenia. Information on the continued efficacy of aripiprazole was also gathered in this long-term trial (until 31 Dec 2012 or until aripiprazole was otherwise available through marketed means and/or reimbursed).

ELIGIBILITY:
Inclusion Criteria:

1. Complete a Prior Study: each patient must meet one of the following conditions for completion of the prior study:

   * A patient who has completed 52 weeks of post-randomization treatment in the prior double blind study (31-97-301 or 31-98-304-01) is eligible, with no further qualifications.
   * A patient who was early-terminated from the study 31-97-301 or 31-98- 304-01 for either of the following two reasons is eligible to enter this open label study with no minimal required duration of prior double-blind participation:

     * Early termination was due to a marked deterioration of clinical status and no serious adverse events (SAE) other than hospitalization has occurred. The marked clinical deterioration must be documented by at least a one-point increase in CGI-Severity score from the baseline and a score of 6 (much worse) or 7 (very much worse) in CGI-Global Improvement at the time of termination, or
     * Early termination was due to a non-serious AE requiring discontinuation of the study drug
   * A patient who was early terminated after a minimum of 4 weeks' participation in the double-blind treatment in study 31-97-301 or 31-98- 304-01 and the reason for early termination was withdrawal of consent due to lack of effect but not marked deterioration. This must be documented by no change from baseline in the CGI-Severity score and a score of 4 (no change) or 5 (minimally worse) on the CGI-Global Improvement scale.
2. Signing of Informed Consent Form: Prior to any procedure or drug administration, each patient must sign an informed consent form. In addition, if required by the Ethical Committee, each patient's next-of-kin or responsible caregiver will co-sign the patient's consent form or a separate consent form.

Exclusion Criteria:

1. Patients suffering from any significant somatic disease or medical problem that would obscure the results of treatment, or that might require frequent changes of concomitant medication.
2. Patients with any acute or unstable medical condition requiring pharmacotherapy, other than schizophrenia.
3. Patients with an abnormal laboratory test value in the most recent analysis (from the study 31-97-301 or 31-98-304-01) which is considered by the investigator as presenting a significant risk to the patient for continuing treatment with aripiprazole.
4. Patients who were early-terminated from the prior double-blind studies (31-97-301 or 31-98-304-01) due to a serious adverse event (SAE) other than worsening of psychosis or hospitalization.
5. Female patients of child bearing potential with a positive serum pregnancy test at the baseline (last visit of prior study) of this open-label follow-on study.
6. Patients who have positive result in the urine screen for drugs of abuse (except for cannabis or medically-prescribed analgesics or benzodiazepines.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 1998-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 631 participants at 139 trial sites in 23 countries.
Pre-assignment Details: All participants enrolled in this trial had previously participated in the double-blind aripiprazole; 89 participants from trial 31-97-301 and 542 participants from trial 31-98-304-01. NCT numbers were not available for these 2 trials as this was before the requirement. Studies were initiated in 1997 (31-97-201) and 1998 (31-98-304-01).
Groups:
- Aripiprazole: All participants began open-label treatment with 30 mg aripiprazole on the first day of participation in the current trial. Once a participant stabilized at the 30 mg per day dose, the study physician could adjust the dose within the range of 10 to 30 mg per day as needed (throughout this long-term trial), to manage adverse events.
Period: Overall Study
Arm/Group | Aripiprazole
Started | 631
Completed | 0
Not Completed | 631
Not completed — Lost to Follow-up | 21
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 236
Not completed — Insufficient Clinical Response | 26
Not completed — Adverse Event | 44
Not completed — Sponsor discontinued trial | 167
Not completed — Noncompliance | 27
Not completed — Protocol Violation | 6
Not completed — Met Withdrawal Criteria | 7
Not completed — AE of Worsening Schizophrenia | 96

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264
  Male | 367

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score by Week
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: All participants who had received at least one dose of study medication were included in both efficacy and safety analyses dataset.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | -1.63 (7.92)
  Week 2 (N= 595) | -3.19 (9.64)
  Week 4 (N= 586) | -4.27 (10.90)
  Week 6 (N= 573) | -4.93 (12.07)
  Week 8 (N= 552) | -5.35 (13.03)
  Week 12 (N= 532) | -5.47 (14.61)
  Week 16 (N= 517) | -6.28 (14.44)
  Week 24 (N= 489) | -6.78 (14.22)
  Week 36 (N= 458) | -7.22 (14.17)
  Week 48 (N= 426) | -8.07 (15.72)
  Week 60 (N= 395) | -9.28 (14.71)
  Week 72 (N= 382) | -9.81 (15.98)
  Week 84 (N= 362) | -10.54 (15.92)
  Week 96 (N= 340) | -10.68 (16.40)
  Week 108 (N= 328) | -11.46 (16.56)
  Week 120 (N= 316) | -11.43 (17.01)
  Week 132 (N= 306) | -11.05 (17.37)
  Week 144 (N= 288) | -11.70 (17.72)
  Week 156 (N= 279) | -11.90 (17.47)
  Week 168 (N= 272) | -11.69 (17.11)
  Week 180 (N= 268) | -11.83 (17.41)
  Week 192 (N= 255) | -11.46 (18.00)
  Week 204 (N= 239) | -12.10 (17.72)
  Week 216 (N= 238) | -11.54 (17.05)
  Week 228 (N= 224) | -12.24 (17.53)
  Week 240 (N= 183) | -12.14 (19.35)
  Week 252 (N= 139) | -15.19 (18.61)
  Week 264 (N= 83) | -22.16 (21.07)
  Week 276 (N= 58) | -29.45 (20.33)
  Week 288 (N= 56) | -28.79 (20.66)
  Week 300 (N= 55) | -21.95 (19.91)
  Week 312 (N= 37) | -25.35 (18.41)
  Week 324 (N= 38) | -21.95 (17.45)
  Week 336 (N= 28) | -24.86 (17.78)
  Week 348 (N= 8) | -12.88 (14.71)
  Week 360 (N= 10) | -17.70 (35.32)
  Week 372 (N= 3) | -10.67 (4.16)
  Week 384 (N= 5) | -4.60 (9.07)
  Week 396 (N= 10) | -10.10 (12.67)
  Week 408 (N= 9) | -5.56 (7.06)
  Week 420 (N= 4) | -8.00 (2.83)
  Week 432 (N= 3) | -13.67 (24.19)
  Week 444 (N= 1) | -28.00 (NA) — Standard deviation (SD) was not calculated as N= 1.
  Week 456 (N= 4) | -48.25 (32.12)
  Week 468 (N= 2) | -36.00 (2.83)
  Week 480 (N= 1) | -10.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -10.00 (13.52)
  Week 504 (N= 2) | -9.50 (28.99)
  Week 636 (N= 5) | -7.60 (22.35)
  Week 648 (N= 2) | -10.00 (14.14)
  Week 660 (N= 3) | -15.33 (19.66)
  Week 672 (N= 1) | 1.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | -7.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | -2.30 (22.21)

2. Primary Outcome: Mean Change From Baseline in PANSS Positive Sub-scale Score by Week
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS Positive Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | -0.39 (2.51)
  Week 2 (N= 595) | -0.81 (3.15)
  Week 4 (N= 586) | -1.13 (3.47)
  Week 6 (N= 573) | -1.23 (3.70)
  Week 8 (N= 552) | -1.30 (3.97)
  Week 12 (N= 533) | -1.24 (4.43)
  Week 16 (N= 517) | -1.43 (4.20)
  Week 24 (N= 489) | -1.54 (4.26)
  Week 36 (N= 458) | -1.56 (4.20)
  Week 48 (N= 426) | -1.73 (4.64)
  Week 60 (N= 395) | -2.01 (4.32)
  Week 72 (N= 382) | -2.08 (4.63)
  Week 84 (N= 362) | -2.26 (4.65)
  Week 96 (N= 340) | -2.26 (4.81)
  Week 108 (N= 328) | -2.50 (4.76)
  Week 120 (N= 316) | -2.45 (4.84)
  Week 132 (N= 306) | -2.25 (5.02)
  Week 144 (N= 289) | -2.49 (5.03)
  Week 156 (N= 279) | -2.46 (4.87)
  Week 168 (N= 272) | -2.35 (4.62)
  Week 180 (N= 268) | -2.40 (4.78)
  Week 192 (N= 255) | -2.22 (4.91)
  Week 204 (N= 239) | -2.48 (4.86)
  Week 216 (N= 238) | -2.21 (4.57)
  Week 228 (N= 224) | -2.42 (4.51)
  Week 240 (N= 183) | -2.10 (5.16)
  Week 252 (N= 139) | -2.74 (4.81)
  Week 264 (N= 83) | -4.24 (5.69)
  Week 276 (N= 58) | -5.90 (5.80)
  Week 288 (N= 56) | -6.30 (5.61)
  Week 300 (N= 55) | -4.16 (5.54)
  Week 312 (N= 37) | -5.27 (5.57)
  Week 324 (N= 38) | -4.45 (5.64)
  Week 336 (N= 28) | -5.46 (5.73)
  Week 348 (N= 8) | -0.75 (1.04)
  Week 360 (N= 10) | -3.80 (7.60)
  Week 372 (N= 3) | -0.67 (0.58)
  Week 384 (N= 5) | -0.80 (3.96)
  Week 396 (N= 10) | -2.40 (3.63)
  Week 408 (N= 9) | -0.89 (2.80)
  Week 420 (N= 4) | -0.75 (1.50)
  Week 432 (N= 3) | -4.67 (8.08)
  Week 444 (N= 1) | -9.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 4) | -10.50 (5.97)
  Week 468 (N= 2) | -6.50 (3.54)
  Week 480 (N= 1) | -2.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -2.00 (2.65)
  Week 504 (N= 2) | -2.50 (7.78)
  Week 636 (N= 5) | -1.80 (4.02)
  Week 648 (N= 2) | -4.50 (7.78)
  Week 660 (N= 3) | -2.00 (2.65)
  Week 672 (N= 1) | 1.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | -1.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | 0.23 (6.58)

3. Primary Outcome: Mean Change From Baseline in PANSS Negative Sub-scale Score by Week
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS Negative Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | -0.35 (2.18)
  Week 2 (N= 595) | -0.82 (2.59)
  Week 4 (N= 586) | -1.05 (3.04)
  Week 6 (N= 573) | -1.24 (3.38)
  Week 8 (N= 552) | -1.41 (3.54)
  Week 12 (N= 532) | -1.54 (4.01)
  Week 16 (N= 517) | -1.85 (4.12)
  Week 24 (N= 489) | -2.02 (4.13)
  Week 36 (N= 458) | -2.16 (4.41)
  Week 48 (N= 426) | -2.43 (4.71)
  Week 60 (N= 395) | -2.75 (4.38)
  Week 72 (N= 382) | -2.94 (4.79)
  Week 84 (N= 362) | -3.17 (4.87)
  Week 96 (N= 340) | -3.22 (4.99)
  Week 108 (N= 328) | -3.36 (4.99)
  Week 120 (N= 316) | -3.37 (5.25)
  Week 132 (N= 306) | -3.41 (5.29)
  Week 144 (N= 288) | -3.58 (5.43)
  Week 156 (N= 279) | -3.70 (5.27)
  Week 168 (N= 272) | -3.68 (5.28)
  Week 180 (N= 268) | -3.69 (5.21)
  Week 192 (N= 255) | -3.65 (5.40)
  Week 204 (N= 239) | -3.79 (5.37)
  Week 216 (N= 238) | -3.74 (5.17)
  Week 228 (N= 224) | -3.90 (5.38)
  Week 240 (N= 183) | -4.09 (5.86)
  Week 252 (N= 139) | -4.88 (5.69)
  Week 264 (N= 83) | -6.87 (6.50)
  Week 276 (N= 58) | -8.71 (6.57)
  Week 288 (N= 56) | -8.32 (6.85)
  Week 300 (N= 55) | -6.58 (6.42)
  Week 312 (N= 37) | -7.51 (5.43)
  Week 324 (N= 38) | -6.63 (4.44)
  Week 336 (N= 28) | -7.43 (4.59)
  Week 348 (N= 8) | -4.88 (5.89)
  Week 360 (N= 10) | -5.60 (9.40)
  Week 372 (N= 3) | -4.33 (1.53)
  Week 384 (N= 5) | 0.00 (2.12)
  Week 396 (N= 10) | -2.90 (3.67)
  Week 408 (N= 9) | -1.22 (2.54)
  Week 420 (N= 4) | -2.25 (2.22)
  Week 432 (N= 3) | -2.67 (7.51)
  Week 444 (N= 1) | -6.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 4) | -13.75 (9.95)
  Week 468 (N= 2) | -9.00 (5.66)
  Week 480 (N= 1) | -5.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -2.00 (3.61)
  Week 504 (N= 2) | -1.50 (12.02)
  Week 636 (N= 5) | -1.80 (5.85)
  Week 648 (N= 2) | 0.00 (0.00)
  Week 660 (N= 3) | -4.67 (6.66)
  Week 672 (N= 1) | 1.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | -3.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | -1.34 (6.09)

4. Primary Outcome: Mean Change From Baseline in Clinical Global Impression of Severity (CGI-S) by Week
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | -0.07 (0.49)
  Week 2 (N= 595) | -0.13 (0.60)
  Week 4 (N= 586) | -0.20 (0.67)
  Week 6 (N= 573) | -0.23 (0.78)
  Week 8 (N= 552) | -0.25 (0.79)
  Week 12 (N= 533) | -0.25 (0.86)
  Week 16 (N= 517) | -0.30 (0.86)
  Week 24 (N= 489) | -0.31 (0.89)
  Week 36 (N= 458) | -0.32 (0.95)
  Week 48 (N= 426) | -0.38 (0.94)
  Week 60 (N= 395) | -0.45 (0.92)
  Week 72 (N= 382) | -0.45 (0.93)
  Week 84 (N= 362) | -0.49 (0.95)
  Week 96 (N= 340) | -0.48 (0.99)
  Week 108 (N= 328) | -0.51 (0.95)
  Week 120 (N= 316) | -0.53 (0.98)
  Week 132 (N= 306) | -0.48 (1.03)
  Week 144 (N= 290) | -0.52 (1.04)
  Week 156 (N= 279) | -0.53 (1.00)
  Week 168 (N= 272) | -0.53 (0.96)
  Week 180 (N= 268) | -0.55 (0.98)
  Week 192 (N= 255) | -0.54 (1.04)
  Week 204 (N= 239) | -0.55 (1.01)
  Week 216 (N= 238) | -0.53 (0.99)
  Week 228 (N= 232) | -0.56 (1.00)
  Week 240 (N= 216) | -0.56 (1.06)
  Week 252 (N= 208) | -0.58 (0.96)
  Week 264 (N= 194) | -0.58 (1.04)
  Week 276 (N= 187) | -0.61 (1.01)
  Week 288 (N= 177) | -0.64 (1.02)
  Week 300 (N= 167) | -0.63 (0.99)
  Week 312 (N= 145) | -0.57 (1.01)
  Week 324 (N= 137) | -0.60 (0.99)
  Week 336 (N= 121) | -0.59 (0.95)
  Week 348 (N= 114) | -0.48 (0.97)
  Week 360 (N= 105) | -0.54 (0.98)
  Week 372 (N= 93) | -0.49 (0.94)
  Week 384 (N= 91) | -0.51 (0.94)
  Week 396 (N= 80) | -0.53 (1.06)
  Week 408 (N= 69) | -0.62 (0.96)
  Week 420 (N= 61) | -0.70 (1.07)
  Week 432 (N= 58) | -0.69 (1.16)
  Week 444 (N= 51) | -0.59 (0.96)
  Week 456 (N= 48) | -0.65 (1.10)
  Week 468 (N= 37) | -0.46 (1.04)
  Week 480 (N= 33) | -0.42 (0.83)
  Week 492 (N= 31) | -0.55 (0.99)
  Week 504 (N= 21) | -0.57 (0.93)
  Week 516 (N= 19) | -0.53 (0.84)
  Week 528 (N= 19) | -0.47 (0.90)
  Week 540 (N= 18) | -0.61 (0.70)
  Week 552 (N= 18) | -0.56 (0.86)
  Week 564 (N= 17) | -0.41 (0.87)
  Week 576 (N= 17) | -0.35 (0.86)
  Week 588 (N= 17) | -0.41 (0.87)
  Week 600 (N= 16) | -0.44 (0.89)
  Week 612 (N= 16) | -0.44 (0.89)
  Week 624 (N= 16) | -0.50 (0.73)
  Week 636 (N= 16) | -0.44 (0.89)
  Week 648 (N= 10) | -0.70 (0.67)
  Week 660 (N= 8) | -0.50 (0.53)
  Week 672 (N= 3) | -0.67 (0.58)
  Week 684 (N= 1) | -1.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | -1.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | -0.00 (1.31)

5. Primary Outcome: Mean Clinical Global Impression of Improvement (CGI-I) by Week
Description: The efficacy of trial medication were rated for each participant using the CGI-I scale. The study physician must rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at baseline. Response choices include: 0 = not assessed; 1 =very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5
  =minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | 3.60 (0.93)
  Week 2 (N= 595) | 3.42 (0.98)
  Week 4 (N= 586) | 3.29 (1.02)
  Week 6 (N= 573) | 3.21 (1.08)
  Week 8 (N= 552) | 3.17 (1.10)
  Week 12 (N= 533) | 3.16 (1.12)
  Week 16 (N= 517) | 3.08 (1.18)
  Week 24 (N= 489) | 3.03 (1.14)
  Week 36 (N= 458) | 2.95 (1.14)
  Week 48 (N= 426) | 2.88 (1.17)
  Week 60 (N= 395) | 2.76 (1.14)
  Week 72 (N= 382) | 2.73 (1.11)
  Week 84 (N= 362) | 2.67 (1.11)
  Week 96 (N= 340) | 2.67 (1.15)
  Week 108 (N= 328) | 2.60 (1.12)
  Week 120 (N= 316) | 2.58 (1.15)
  Week 132 (N= 306) | 2.62 (1.17)
  Week 144 (N= 290) | 2.59 (1.20)
  Week 156 (N= 279) | 2.58 (1.16)
  Week 168 (N= 272) | 2.57 (1.15)
  Week 180 (N= 268) | 2.57 (1.16)
  Week 192 (N= 255) | 2.59 (1.20)
  Week 204 (N= 239) | 2.56 (1.16)
  Week 216 (N= 238) | 2.56 (1.20)
  Week 228 (N= 232) | 2.49 (1.17)
  Week 240 (N= 216) | 2.48 (1.21)
  Week 252 (N= 208) | 2.37 (1.13)
  Week 264 (N= 194) | 2.14 (1.07)
  Week 276 (N= 187) | 2.16 (1.03)
  Week 288 (N= 177) | 2.26 (1.06)
  Week 300 (N= 167) | 2.26 (1.16)
  Week 312 (N= 145) | 2.18 (1.11)
  Week 324 (N= 137) | 2.23 (1.05)
  Week 336 (N= 121) | 2.03 (1.09)
  Week 348 (N= 114) | 2.45 (1.00)
  Week 360 (N= 105) | 2.53 (1.36)
  Week 372 (N= 93) | 2.14 (1.07)
  Week 384 (N= 91) | 2.50 (1.52)
  Week 396 (N= 80) | 3.00 (1.63)
  Week 408 (N= 69) | 2.50 (1.18)
  Week 420 (N= 61) | 2.43 (1.40)
  Week 432 (N= 58) | 2.00 (1.73)
  Week 444 (N= 51) | 1.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 48) | 1.83 (0.75)
  Week 468 (N= 37) | 2.00 (0.00)
  Week 480 (N= 33) | 2.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | 2.33 (1.32)
  Week 504 (N= 2) | 2.50 (2.12)
  Week 528 (N= 1) | 4.00 (NA) — SD was not calculated as N= 1.
  Week 636 (N= 5) | 2.00 (0.00)
  Week 648 (N= 2) | 1.50 (0.71)
  Week 660 (N= 3) | 2.33 (1.15)
  Week 672 (N= 3) | 1.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | 1.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | 3.35 (1.60)

6. Primary Outcome: Mean Change From Baseline in Montgomery and Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in participants with mood disorders. The questionnaire includes questions on the following symptoms. 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The usual cut-off points are: 0 to 6 = normal/ symptom absent, 7 to 19 = mild depression, 20 to 34 = moderate depression, >34 = severe depression.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | -0.78 (3.62)
  Week 2 (N= 595) | -1.13 (4.09)
  Week 4 (N= 586) | -1.38 (4.73)
  Week 6 (N= 572) | -1.54 (5.15)
  Week 8 (N= 552) | -1.40 (4.98)
  Week 12 (N= 533) | -1.31 (5.77)
  Week 16 (N= 517) | -1.60 (5.41)
  Week 24 (N= 489) | -1.61 (5.75)
  Week 36 (N= 458) | -1.66 (5.75)
  Week 48 (N= 425) | -1.75 (5.47)
  Week 60 (N= 395) | -2.13 (5.41)
  Week 72 (N= 382) | -2.21 (5.29)
  Week 84 (N= 362) | -2.33 (5.51)
  Week 96 (N= 339) | -2.26 (5.70)
  Week 108 (N= 328) | -2.30 (5.68)
  Week 120 (N= 316) | -2.40 (5.67)
  Week 132 (N= 306) | -2.22 (5.85)
  Week 144 (N= 291) | -2.47 (5.85)
  Week 156 (N= 279) | -2.51 (5.64)
  Week 168 (N= 272) | -2.51 (5.49)
  Week 180 (N= 268) | -2.73 (5.67)
  Week 192 (N= 255) | -2.53 (6.05)
  Week 204 (N= 239) | -2.69 (6.20)
  Week 216 (N= 238) | -2.50 (5.87)
  Week 228 (N= 224) | -2.62 (5.82)
  Week 240 (N= 183) | -2.92 (6.50)
  Week 252 (N= 139) | -3.63 (6.53)
  Week 264 (N= 83) | -5.52 (7.89)
  Week 276 (N= 58) | -7.71 (8.88)
  Week 288 (N= 56) | -7.57 (8.64)
  Week 300 (N= 55) | -6.15 (7.52)
  Week 312 (N= 37) | -7.24 (8.51)
  Week 324 (N= 38) | -6.32 (8.76)
  Week 336 (N= 28) | -7.21 (8.01)
  Week 348 (N= 8) | -4.00 (7.45)
  Week 360 (N= 10) | -2.80 (16.09)
  Week 372 (N= 3) | -2.67 (2.08)
  Week 384 (N= 5) | 0.00 (0.00)
  Week 396 (N= 10) | -1.40 (2.95)
  Week 408 (N= 9) | -1.89 (1.27)
  Week 420 (N= 4) | 0.75 (4.11)
  Week 432 (N= 3) | -2.33 (5.86)
  Week 444 (N= 1) | -1.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 5) | -9.60 (8.85)
  Week 468 (N= 2) | -3.00 (2.83)
  Week 480 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -6.56 (8.44)
  Week 504 (N= 2) | -13.50 (13.44)
  Week 636 (N= 5) | 0.40 (3.36)
  Week 648 (N= 2) | -1.00 (1.41)
  Week 660 (N= 3) | -4.33 (2.31)
  Week 672 (N= 1) | -2.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | -1.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | -0.31 (8.02)

7. Primary Outcome: Mean Change From Baseline in Simpson-Angus Scale (SAS) Total Score by Week
Description: The SAS is composed of 10 items. This scale contains 10 items: Gait, Arm dropping, Shoulder shaking, Elbow rigidity, Wrist rigidity, Head rotation, Glabella Tap, Tremor, Salivation, Akathisia. Grade of severity of each item is rated using a 5-point scale, 1 (normal) and 5 (most severe). The total score ranges from 10 to 50. Negative changes from baseline indicate an improvement, with higher negative values indicating better improvement.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 618) | -0.78 (3.05)
  Week 2 (N= 594) | -1.01 (3.32)
  Week 4 (N= 585) | -1.06 (3.68)
  Week 6 (N= 572) | -1.14 (3.94)
  Week 8 (N= 550) | -1.19 (4.00)
  Week 12 (N= 532) | -1.28 (4.03)
  Week 16 (N= 516) | -1.27 (4.18)
  Week 24 (N= 488) | -1.24 (3.91)
  Week 36 (N= 456) | -1.10 (3.79)
  Week 48 (N= 426) | -1.33 (4.14)
  Week 60 (N= 395) | -1.25 (3.89)
  Week 72 (N= 382) | -1.36 (4.07)
  Week 84 (N= 362) | -1.33 (4.16)
  Week 96 (N= 338) | -1.24 (3.92)
  Week 108 (N= 328) | -1.29 (3.83)
  Week 120 (N= 316) | -1.22 (3.83)
  Week 132 (N= 306) | -1.26 (3.88)
  Week 144 (N= 289) | -1.26 (3.99)
  Week 156 (N= 278) | -1.33 (4.04)
  Week 168 (N= 272) | -1.31 (3.92)
  Week 180 (N= 268) | -1.43 (4.08)
  Week 192 (N= 255) | -1.46 (4.07)
  Week 204 (N= 239) | -1.49 (4.16)
  Week 216 (N= 238) | -1.39 (3.48)
  Week 228 (N= 224) | -1.44 (3.55)
  Week 240 (N= 183) | -1.68 (3.72)
  Week 252 (N= 139) | -2.11 (4.16)
  Week 264 (N= 83) | -2.89 (4.99)
  Week 276 (N= 58) | -3.84 (5.64)
  Week 288 (N= 56) | -3.88 (5.77)
  Week 300 (N= 55) | -2.53 (4.55)
  Week 312 (N= 37) | -2.30 (4.07)
  Week 324 (N= 38) | -1.76 (4.10)
  Week 336 (N= 28) | -1.64 (3.90)
  Week 348 (N= 8) | -2.00 (2.78)
  Week 360 (N= 9) | -0.44 (5.75)
  Week 372 (N= 3) | -1.00 (0.00)
  Week 384 (N= 5) | -0.20 (0.45)
  Week 396 (N= 10) | -0.30 (1.16)
  Week 408 (N= 9) | -0.89 (1.27)
  Week 420 (N= 4) | -1.25 (1.50)
  Week 432 (N= 3) | -1.00 (1.73)
  Week 444 (N= 1) | 1.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 5) | -7.20 (8.87)
  Week 468 (N= 2) | 0.00 (0.00)
  Week 480 (N= 1) | -1.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -3.22 (5.33)
  Week 504 (N= 2) | -3.00 (4.24)
  Week 636 (N= 5) | -0.20 (0.45)
  Week 648 (N= 2) | 0.00 (0.00)
  Week 660 (N= 3) | -1.00 (1.00)
  Week 672 (N= 1) | -3.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | -7.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 628) | -1.36 (4.31)

8. Primary Outcome: Mean Change From Baseline in Barnes Akathisia Rating Scale Score (BARS) Total Score by Week
Description: BARS consisted of 4 items: objective observation of akathisia by study physician, subjective feelings of restlessness by participant, participant distress due to akathisia, global evaluation of akathisia. The first 3 items were rated on a 4-point scale: 0 = absence of symptoms to 3 = severe condition. The global clinical evaluation were made on a 6-point scale, (0=absent, 1=questionable, 2=mild, 3=moderate, 4=marked, 5=severe). Participants were observed while they were seated and then stood for a minimum of 2 minutes in each position. Symptoms observed in other situations (e.g., while engaged in neutral conversation or engaged in activity on the ward) may also be rated. Subjective phenomena were elicited by direct questioning. The BARS Global Score was derived from the global clinical assessment of akathisia from the BARS panel. Total score ranges from 0 to 14. Negative changes from baseline indicate improvement, with higher negative values indicating better improvement.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 618) | -0.15 (0.67)
  Week 2 (N= 595) | -0.20 (0.70)
  Week 4 (N= 586) | -0.20 (0.74)
  Week 6 (N= 572) | -0.23 (0.76)
  Week 8 (N= 552) | -0.22 (0.79)
  Week 12 (N= 533) | -0.22 (0.78)
  Week 16 (N= 517) | -0.22 (0.77)
  Week 24 (N= 489) | -0.22 (0.74)
  Week 36 (N= 458) | -0.21 (0.75)
  Week 48 (N= 425) | -0.20 (0.75)
  Week 60 (N= 395) | -0.20 (0.70)
  Week 72 (N= 382) | -0.19 (0.73)
  Week 84 (N= 362) | -0.21 (0.74)
  Week 96 (N= 340) | -0.21 (0.79)
  Week 108 (N= 327) | -0.21 (0.77)
  Week 120 (N= 316) | -0.20 (0.75)
  Week 132 (N= 306) | -0.22 (0.76)
  Week 144 (N= 291) | -0.22 (0.79)
  Week 156 (N= 278) | -0.24 (0.79)
  Week 168 (N= 272) | -0.22 (0.78)
  Week 180 (N= 268) | -0.24 (0.81)
  Week 192 (N= 255) | -0.29 (0.79)
  Week 204 (N= 238) | -0.29 (0.80)
  Week 216 (N= 237) | -0.26 (0.76)
  Week 228 (N= 223) | -0.26 (0.78)
  Week 240 (N= 183) | -0.24 (0.75)
  Week 252 (N= 139) | -0.29 (0.81)
  Week 264 (N= 83) | -0.51 (1.06)
  Week 276 (N= 58) | -0.69 (1.16)
  Week 288 (N= 56) | -0.64 (1.09)
  Week 300 (N= 55) | -0.51 (0.96)
  Week 312 (N= 37) | -0.35 (0.68)
  Week 324 (N= 38) | -0.26 (0.60)
  Week 336 (N= 28) | -0.29 (0.66)
  Week 348 (N= 8) | -0.75 (1.04)
  Week 360 (N= 9) | -0.22 (0.67)
  Week 372 (N= 3) | 0.00 (0.00)
  Week 384 (N= 5) | 0.00 (0.00)
  Week 396 (N= 10) | -0.10 (0.32)
  Week 408 (N= 9) | -0.33 (0.71)
  Week 420 (N= 4) | -0.25 (0.50)
  Week 432 (N= 3) | 0.00 (0.00)
  Week 444 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 5) | -1.40 (1.67)
  Week 468 (N= 2) | 0.00 (0.00)
  Week 480 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -0.56 (1.01)
  Week 504 (N= 2) | -1.50 (0.71)
  Week 636 (N= 5) | -0.40 (0.89)
  Week 648 (N= 2) | 0.00 (0.00)
  Week 660 (N= 3) | -0.67 (1.15)
  Week 672 (N= 1) | -4.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | -0.26 (0.85)

9. Primary Outcome: Mean Change From Baseline in Abnormal Involuntary Movement Scale Score (AIMS) Total Score by Week
Description: The AIMS assessment consisted of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) were observed unobtrusively while the participant was at rest (e.g., in the waiting room), and the study physician would make global judgments on the participant's dyskinesia's (items 8 through 10). For this scale, the participant was seated on a hard, firm chair. These items are rated on a five-point scale: 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). The total score ranges from 0 to 40. Negative changes from baseline indicate an improvement, with higher negative values indicating better improvement.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Units on a scale
  Week 1 (N= 619) | -0.21 (1.61)
  Week 2 (N= 595) | -0.29 (1.77)
  Week 4 (N= 586) | -0.28 (1.96)
  Week 6 (N= 572) | -0.34 (2.25)
  Week 8 (N= 552) | -0.34 (2.22)
  Week 12 (N= 533) | -0.37 (2.26)
  Week 16 (N= 517) | -0.39 (2.31)
  Week 24 (N= 489) | -0.35 (2.08)
  Week 36 (N= 458) | -0.21 (1.85)
  Week 48 (N= 425) | -0.35 (2.17)
  Week 60 (N= 395) | -0.33 (2.02)
  Week 72 (N= 382) | -0.31 (2.10)
  Week 84 (N= 362) | -0.31 (2.12)
  Week 96 (N= 340) | -0.25 (1.84)
  Week 108 (N= 328) | -0.27 (1.88)
  Week 120 (N= 316) | -0.26 (1.85)
  Week 132 (N= 306) | -0.26 (1.91)
  Week 144 (N= 290) | -0.29 (1.97)
  Week 156 (N= 279) | -0.31 (2.04)
  Week 168 (N= 272) | -0.29 (1.87)
  Week 180 (N= 268) | -0.34 (2.08)
  Week 192 (N= 255) | -0.35 (2.08)
  Week 204 (N= 239) | -0.30 (2.06)
  Week 216 (N= 238) | -0.26 (1.50)
  Week 228 (N= 224) | -0.31 (1.41)
  Week 240 (N= 183) | -0.31 (1.44)
  Week 252 (N= 139) | -0.40 (1.59)
  Week 264 (N= 83) | -0.61 (1.95)
  Week 276 (N= 58) | -0.76 (2.30)
  Week 288 (N= 56) | -0.57 (2.72)
  Week 300 (N= 55) | -0.18 (1.45)
  Week 312 (N= 37) | -0.35 (0.68)
  Week 324 (N= 38) | -0.32 (0.57)
  Week 336 (N= 28) | -0.36 (0.56)
  Week 348 (N= 8) | -0.50 (1.07)
  Week 360 (N= 9) | -0.44 (0.73)
  Week 372 (N= 3) | 0.00 (0.00)
  Week 384 (N= 5) | 0.00 (0.00)
  Week 396 (N= 10) | 0.00 (0.00)
  Week 408 (N= 9) | 0.00 (0.00)
  Week 420 (N= 4) | 0.00 (0.00)
  Week 432 (N= 3) | 0.00 (0.00)
  Week 444 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Week 456 (N= 5) | -1.00 (2.24)
  Week 468 (N= 2) | 0.00 (0.00)
  Week 480 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Week 492 (N= 9) | -0.44 (0.53)
  Week 504 (N= 2) | -0.50 (0.71)
  Week 636 (N= 5) | 0.20 (0.45)
  Week 648 (N= 2) | 0.00 (0.00)
  Week 660 (N= 3) | 0.00 (0.00)
  Week 672 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Week 696 (N= 1) | 0.00 (NA) — SD was not calculated as N= 1.
  Last Visit (N= 629) | -0.39 (2.36)

10. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The AEs were one of the primary parameters to measure the safety and tolerability of individual participants. The AEs were captured for all participants from the time the ICF was signed until the end of the trial.
Time Frame: Baseline to Last Visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Participants
  Participants with serious TEAEs | 179
  Participants with severe TEAEs | 116
  Participants discontinued medication due to AE | 140
  Participants with TEAEs | 523
  Participants discontinued due to AEs or death | 140

11. Primary Outcome: Percentage of Participants With Vital Signs of Potential Clinical Relevance
Description: The vital signs were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance included abnormal values in heart rate, systolic and diastolic blood pressure, respiratory rate and weight that were identified based on pre-defined criteria.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
percentage of participants
  Heart rate sitting increase ≥15 bpm (N=625) | 0.5
  Systolic sitting BP increase ≥20 mmHg (N=627) | 0.8
  Systolic sitting BP decrease ≥20 mmHg (N=627) | 1.3
  Diastolic sitting BP increase ≥15mmHg (N=627) | 3.0
  Weight gain ≥7% (N=622) | 38.9
  Weight loss ≥7% (N=622) | 23.6

12. Primary Outcome: Percentage of Participants With ECG Measurements of Potential Clinical Relevance
Description: The measurement of ECG was one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, QRS, QT, QTcB, and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Percentage of participants
  Tachycardia (N=612) | 0.8
  Bradycardia (N=612) | 7.5
  Sinus tachycardia (N=612) | 0.8
  Sinus bradycardia (N=612) | 7.4
  Ventricular premature beat (N=612) | 2.9
  Primary atrioventricular block (N=606) | 2.5
  Secondary atrioventricular block (N=612) | 0.2
  Left bundle branch block (N=612) | 0.2
  Right bundle branch block (N=612) | 16.0
  Pre-excitation syndrome (N=612) | 0.3
  Other intraventricular conduction block (N=611) | 1.8
  Acute infarction (N=612) | 0.2
  Old infarction (N=612) | 0.7
  QTcB (N=612) | 8.0
  QTcF (N=611) | 2.1
  QTcN (N=611) | 2.3

13. Primary Outcome: Percentage of Participants With Laboratory Values of Potential Clinical Relevance
Description: The laboratory values were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, 108 continuing every 12 weeks, Last Visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 631
Percentage of participants
  Alanine aminotransferase (IU/L) (N=626) | 1.1
  Aspartate aminotransferase (IU/L) (N=626) | 1.0
  Bilirubin (mg/dl) (high)(N=626) | 3.0
  Calcium (mg/dl) (low) (N=626) | 3.4
  Chloride (meq/l) (low) (N=626) | 0.5
  Chloride (meq/l) (high) (N=626) | 0.2
  Creatinine phosphokinase (IU/L) (N=626) | 14.9
  Creatinine (mg/dl) (N=617) | 0.5
  Glucose (mg/dl) (N=626) | 3.0
  Lactic dehydrogenase (IU/L) (N=626) | 0.2
  Potassium (meq/l) (low) (N=626) | 0.2
  Potassium (meq/l) (high) (N=626) | 5.3
  Sodium (meq/l) (low) (N=626) | 0.5
  Sodium (meq/l) (high) (N=626) | 0.2
  Urea nitrogen (mg/dl) (N=626) | 0.8
  Uric acid (mg/dl) (N=626) | 1.0
  Eosinophils (%) (N=624) | 3.2
  Hematocrit (%) (N=623) | 2.7
  Hemoglobin (g/dl) (N=625) | 2.4
  Platelet count (per cubic mm) (low) (N=625) | 0.2
  Platelet count (per cubic mm) (high) (N=625) | 0.3
  White blood count (thou/mcl) (low) (N=625) | 1.1
  White blood count (thou/mcl) (high) (N=625) | 3.8
  Glucose, urine (N=613) | 1.6
  Protein, urine (N=599) | 1.8

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent to 30 days after the end of study treatment. The investigator continued to report any significant follow-up information on the AE up to the time the event had been resolved.
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 179/631
Other Adverse Events (participants affected / at risk) | 364/631
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=631)
Anemia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 2
Traumatic liver injury (Injury, poisoning and procedural complications) | 1
Blood creatinine phosphokinase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Musculoskeletal and connective tissue disorders) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Akathisia (Nervous system disorders) | 2
Carpal tunnel syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 2
Adjustment disorder (Psychiatric disorders) | 1
Agression (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 2
Alcohol abuse (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 10
Completed suicide (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Depressive symptom (Psychiatric disorders) | 1
Drug abuse (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 4
Hypomania (Psychiatric disorders) | 1
Illusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Persecutory delusion (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 20
Restlessness (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 85
Schizophrenia, paranoid type (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Suicidal attempt (Psychiatric disorders) | 6
Bartholin's cyst (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Prostatic disorder (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Homicide (Social circumstances) | 1
Respite care (Social circumstances) | 2
Social stay hospitalisation (Social circumstances) | 16
Substance use (Social circumstances) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=631)
Influenza (Infections and infestations) | 47
Weight increased (Investigations) | 56
Akathisia (Nervous system disorders) | 84
Extrapyramidal disorder (Nervous system disorders) | 50
Headache (Nervous system disorders) | 48
Tremor (Nervous system disorders) | 50
Anxiety (Psychiatric disorders) | 73
Insomnia (Psychiatric disorders) | 118
Schizophrenia (Psychiatric disorders) | 79

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the sponsor. The protocol specified that the study would run until Abilify (aripiprazole) was commercially available in all site countries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No